CLINICAL TRIAL: NCT01514422
Title: Minocycline for Bipolar Disorder
Brief Title: Minocycline for Bipolar Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Dan V. Iosifescu, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 11-0432
Record Dates: First submitted 2012-01-10; First posted 2012-01-23 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Bipolar Depression
Keywords: Bipolar disorder; depression; minocycline; mood disorders; bipolar depression
MeSH Terms: conditions — Bipolar Disorder; Depression; cyclopia sequence; Mood Disorders | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Minocycline (Experimental): All subjects will be given minocycline over 8 weeks
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Minocycline 100 to 300mg per day for 8 weeks
  Other Names: Minocin

SUMMARY:
The purpose of this study is to evaluate minocycline as a potential treatment for bipolar depression when added to a mood-stabilizing medication. Minocycline is an antibiotic that is approved for the treatment of infections and acne. Participation in this research study is expected to last 8 weeks, and includes five outpatient visits.

DETAILED DESCRIPTION:
Bipolar depression remains the great unmet need in the treatment of bipolar disorder. Only two treatments have been FDA-approved for the management of acute bipolar depression (the combination of olanzapine and fluoxetine and quetiapine). Early pilot data suggests the drug minocycline has potent antidepressant effects. Minocycline is approved by the Food and Drug Administration (FDA) (for acne and bacterial infections), is inexpensive and readily available in generic formulation, and is generally well-tolerated. This study will examine whether administering the drug minocycline to individuals with bipolar depression over 8 weeks will improve their depressive symptoms. This study will also offer an option to participate in proton magnetic resonance spectroscopy (1H-MRS) to measure N-Acetylaspartate (NAA) levels in the brain, which are thought to be decreased in bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for Bipolar I Disorder or Bipolar II disorder, depressed phase
* A baseline score of at least 18 on the Montgomery-Asberg Depression Rating Scale (MADRS)
* Participants on mood stabilizer medication for at least two weeks prior to starting the study, and must remain on the treatment during the study
* Able to understand English

Exclusion Criteria:

* DSM-IV diagnosis of Bipolar NOS, Cyclothymia, or Schizoaffective Bipolar type
* Pregnant women or women of child bearing potential who are not using a medically accepted means of contraception (defined as oral contraceptive pill or implant, condom, diaphragm, spermicide, IUD, s/p tubal ligation, partner with vasectomy)
* Serious suicide or homicide risk
* Unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease
* Clinical or laboratory evidence of hypothyroidism; if maintained on thyroid medication must be euthyroid for at least 1 month before visit 1
* Drug/alcohol dependence within past 30 days, or current substance use disorder that requires detoxification
* Current use of minocycline or history of anaphylactic reaction or intolerance to minocycline
* Primary clinical diagnosis of antisocial or borderline personality disorder
* Patients with metallic foreign bodies or claustrophobia will be excluded from the MRS component

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan V Iosifescu, MD, MSc, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study procedures were conducted between June 2011 and June 2013 at the Mood and Anxiety Disorders Program at Icahn School of Medicine at Mount Sinai.
Period: Overall Study
Arm/Group | Minocycline
Started | 20
Completed | 19
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Minocycline
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (12.7)
Gender [Count of Participants; unit: Participants]
  Female | 8
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Scores on the Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Measured at baseline and week 8. The MADRS-S has 10-items which are based on mood symptoms over the past 7 days. Each items is scored 0 (normal) to 6 (severe depression) with overall score ranges from 0 (normal) to 60 (severe depression).
Time Frame: baseline and week 8
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Minocycline: Minocycline for 8 weeks
Arm/Group | Minocycline
Number analyzed (Participants) | 19
units on a scale | -14.6 [-21.3 to -7.8]

2. Secondary Outcome: Change in N-acetylaspartate (NAA), as Measured by 1H-MRS Scan
Description: Measured at baseline and week 8
Time Frame: baseline and week 8
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Minocycline
Number analyzed (Participants) | 19
mmol/L | 0.001 (0.0022)

3. Secondary Outcome: Changes in Young Mania Rating Scale (YMRS)
Description: Measured at baseline and week 8. The YMRS is an 11-item questionnaire to measure the severity of manic symptoms. 7 items are scored 0-4 and the other 4 items are scored 0-8, with overall score range from 0 (normal) to 60 (severe mania).
Time Frame: baseline and week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Minocycline
Number analyzed (Participants) | 19
units on a scale
  baseline | 1.8 (2.3)
  week 8 | 1.1 (0.9)

ADVERSE EVENTS:
Arm/Group | Minocycline
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Minocycline (N=20)
Frequent need to urinate (Renal and urinary disorders) | 5
Trouble sleeping (General disorders) | 4
Fee!ing drowsy or sleepy (General disorders) | 4
Dry mouth (Skin and subcutaneous tissue disorders) | 4
Muscle cramps or stiffness (Musculoskeletal and connective tissue disorders) | 4
Diarrhea (Gastrointestinal disorders) | 4
Appetite increased (Gastrointestinal disorders) | 4
Difficulties finding words (Nervous system disorders) | 4
Feeling nervous or hyper (Psychiatric disorders) | 3
Irritable (General disorders) | 3
Feeling strange or unreal (Psychiatric disorders) | 3
Stomach or abdominal discomfort (Gastrointestinal disorders) | 3
Difficulty starting urination (Renal and urinary disorders) | 3
Weight gain (General disorders) | 3
Nightmares or other disturbances (Psychiatric disorders) | 2
Weakness or fatigue (Psychiatric disorders) | 2
Dizziness or faintness (Nervous system disorders) | 2
Drooling or increase salivation (Nervous system disorders) | 2
Nausea or vomiting (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Problems with sexual arousal (Psychiatric disorders) | 2
Delayed or absent orgasm (Psychiatric disorders) | 2
Appetite decreased (Gastrointestinal disorders) | 2
Skin rash or allergy (Skin and subcutaneous tissue disorders) | 2
Diminished mental acuity (Psychiatric disorders) | 2
Apathy/emotional indifference (Psychiatric disorders) | 2
Bruising (Blood and lymphatic system disorders) | 2
Hot flashes (Endocrine disorders) | 2
Strange taste in mouth (General disorders) | 2
Unable to sit still (General disorders) | 2
Function impairment (General disorders) | 2

LIMITATIONS AND CAVEATS:
Limitations are this is an open label study with no placebo and low number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes